# Effect of alternating pressure overlay on weight bearing tissue tolerance in people with SCI

#### **Principal Investigator:**

Yi-Ting Tzen, Department of Physical Therapy, UIC; 1919 West Taylor St. Rm 506H, Chicago IL 60612; (312) 996-1506; <a href="mailto:tzenyt@uic.edu">tzenyt@uic.edu</a>

**Study Location(s):** University of Illinois at Chicago, Applied Health Sciences Building, 1919 W Taylor St., room 272, Chicago IL 60612

Sponsor: Dabir Surfaces Inc.

Version: 2

**Date:** April 4, 2017

#### **TABLE OF CONTENTS**

| | Page |
|------------------------------------------------------------|------|
| Table of Contents | |
| List of Abbreviations | |
| 1.0 Project Summary/Abstract | |
| 2.0 Background/Scientific Rationale | |
| 3.0 Objectives/Aims | 6 |
| 4.0 Eligibility | |
| 4.1 Inclusion Criteria | |
| 4.2 Exclusion Criteria | |
| 4.3 Excluded or Vulnerable Populations | 7 |
| 5.0 Subject Enrollment | 8 |
| 6.0 Study Design and Procedures | 9 |
| 7.0 Expected Risks/Benefits | 11 |
| 8.0 Data Collection and Management Procedures | |
| 9.0 Data Analysis | 14 |
| 10.0 Quality Control and Quality Assurance | |
| 11.0 Data and Safety Monitoring | |
| 12.0 Statistical Considerations | |
| 13.0 Regulatory Requirements | |
| 13.1 Informed Consent | |
| 13.2 Subject Confidentiality | 16 |
| 13.3 Unanticipated Problems | 17 |
| 14.0 References | 18 |
| Appendices | 19 |
| American Spinal Injury Association (ASIA) Impairment Scale | 19 |
| Form A: confidential info | 20 |
| Form B: Demographic Info | 21 |
| Form C1 – Self-report Medical History | 22 |
| Form C2 – Self-report CURRENT MEDICATION | 23 |
| Form D – Self-report SOcial HIstory | |
| Form E1 – resting vitals | |
| Form E2 – ASIA Impairment Scale | |
| Form E3 – Autonomic function scale | |
| FORM F – Test Data | |
| FORM G – Compensation | 30 |

#### **LIST OF ABBREVIATIONS**

AIS American Spinal Injury Association Impairment Scale

AP Alternating Pressure

ASIA American Spinal Injury Association

ATP Adenosine Tri Phosphate

CTRL Control

FDA Food and Drug Administration

HH Heat Hyperemic

IRB Institutional Review Board

ISCOS International Spinal Cord Society

LDF Laser Doppler Flowmetry

OR Operation Room
PI Principal Investigator
RH Reactive Hyperemic
ROM Range Of Motion
SBF Skin Blood Flow
SCI Spinal Cord Injury

STFT Short Time Fourier Transform

WLRS White Light Reflectance Spectroscopy

#### 1.0 Project Summary/Abstract

Tissue ischemia (lack of blood flow) is one of the main causes of pressure injury. It is inevitable during bed-ridden condition or prolonged surgery procedure in the operating room. Previous studies demonstrated that the protective mechanisms of alternating pressure (AP) on pressure injury include redistribution of surface pressure, and allowing more blood supplies while lying on the support surface. The Dabir AP overlay is low profile yet possesses similar characteristics as other AP mattresses on the market. The objective of this study is to evaluate the protective mechanisms of Dabir AP overlay on weight bearing tissue of people with chronic spinal cord injury (SCI). Our central hypothesis is that the Dabir AP overlay will cause lower amount of interface pressure and allow more skin blood flow during weight bearing as compared to regular operation room (OR) overlay. In addition, people with SCI will have better tolerance to prolonged weight bearing after preconditioned with the Dabir AP overlay. This study will be repeated measures design, with subjects acting as their own control. Fifteen adults with chronic SCI will be recruited from the Greater Chicago area. Each subject will undergo two study protocols: lying on AP overlay followed by OR overlay (40 minutes each), and lying on OR overlay for 40 minutes only. Laser Doppler flowmetry system will be used to collect data before during and after lying on the overlays, and pressure mapping system will be used to measure interface pressure. Paired *t*-tests will be computed to compare the interface pressure and skin blood flow before, during and after lying on the overlays. Findings of this study will help determine the effectiveness of the Dabir AP overlay on pressure redistribution and ischemia preconditioning.

#### 2.0 Background/Scientific Rationale

Tissue ischemia is one of the main etiologies of pressure injury. It is inevitable during bed-ridden and wheelchair bound conditions, such as spinal cord injury (SCI), or prolonged surgery procedure in the operating room. Active alternating pressure (AP) mattresses are covered by Medicare policy for patients with multiple/large stage 2/ stage 3 pressure injuries to relief interface pressure and prevent recurrence of pressure injuries. Previous studies demonstrated that the protective mechanisms of AP on pressure injury include redistribution of surface pressure, and allowing more blood supplies while lying on the support surface. The Dabir AP overlay (DabirAIR<sup>TM</sup>, Dabir Surfaces Inc., Hardwood Heights, IL) is low profile yet possesses similar characteristics as other AP mattresses on the market; it is intended for clinical use, such as operation room (OR) where AP mattresses may not be an option. We expect Dabir AP overlay will be beneficial to people at risk of pressure injury by maintaining the blood supply during weight bearing condition.

In addition to pressure redistribution and increasing blood supplies, we also postulate that the if an AP overlay will be beneficial to the weight-bearing skin by means of preconditioning the skin with short-term ischemia, i.e. when air cells inflate. Ischemic preconditioning is a method used to prevent tissue damage caused by ischemic events, such as stroke and myocardial infarction, by means of slowing down ATP depletion in the short-term subsequent ischemic episodes and washing out the harmful catabolites during each short-term period of reperfusion. Recently, this method is implemented to heal diabetic foot ulcer by remotely precondition the lower limb. We hypothesize that the alternating pressure characteristics of the Dabir AP overlay could be utilized as a method for preconditioning to protect weight-bearing tissue in people with SCI.

To quantify the severity of tissue ischemia, we will collect the non-invasive reactive hyperemic response as an outcome. Reactive hyperemia is characterized by sudden increase in blood flow after temporary obstruction of the blood flow. Previous studies used this response to simulate the tissue response toward ischemia in people that are at risk of pressure ulcer, such as spinal cord injury.<sup>8,9</sup>

People with SCI are at extremely high risk of pressure ulcer formation due to immobility and lack of sensation. In addition, this population may also have underlying change in vascular control mechanisms. To further quantify the vascular control mechanisms in our participants, we plan to use two additional protocols to provide objective measurements of blood supplies. The two non-invasive measurements are heat hyperemia and skin vasomotor response.

Heat hyperemia is an objective and non-invasive method to quantify the degree of impaired thermoregulation. It is characterized by a biphasic pattern with an initial peak (initiated by activity of sensory nerves and modulated by sympathetic nerves), followed by a brief nadir and a plateau phase (mediated by local production of endothelial nitric oxide).<sup>8</sup> A previous study showed that the initial peak was diminished significantly at skin sites below level of injury in patients with complete SCI.<sup>9</sup> Given that increased skin temperature is a well-proven risk factor in ulcer formation in addition to prolonged pressure, <sup>10</sup> adopting measurement of thermoregulatory function may assist in understanding the pathological patterns related to ulcer formation.

Skin vasomotor response is a reduction in SBF induced by standardized cutaneous electrical stimulation. It is an objective method to assess the integrity of sympathetic pathways, 11 and it is a sensitive tool in identifying sympathetic function below a spinal cord lesion. 12 Measurement of the skin vasomotor response may provide us a comprehensive understanding of the changes in control mechanisms with the pathological pattern in SBF detected before ulcer formation.

By comparing the skin blood flow responses between using Dabir AP overlay vs. standard OR overlay, we might be able to fill the gap of current research by determining the potential benefit of Dabir AP overlay on pressure ulcer prevention.

#### 3.0 Objectives/Aims

The <u>objective</u> of this study is to evaluate the protective mechanisms of Dabir AP overlay on weight bearing tissue of people with chronic spinal cord injury (SCI). Our central hypothesis is that the Dabir AP overlay will cause lower amount of interface pressure and allow more skin blood flow during weight bearing as compared to regular OR overlay. In addition, people with SCI will have better tolerance to prolonged weight bearing after preconditioned with the Dabir AP overlay.

There are three aims (with related hypotheses) for this study:

Aim 1: To determine the effectiveness of pressure redistribution with Dabir AP overlay.

**Hypothesis 1.** Our participants will demonstrate lower interface pressure at sacrum and heel when lying supine for 40 minutes on Dabir AP overlay as compared to that on regular OR overlay (AliMed®).

Aim 2: To examine the severity of tissue ischemia with the use of Dabir AP overlay.

**Hypothesis 2a.** Our participants will demonstrate greater skin blood flow at sacrum and heel when lying supine for 40 minutes on Dabir AP overlay as compared to that on regular OR overlay.

**Hypothesis 1b.** Our participants will demonstrate smaller reactive hyperemic response at sacrum and heel after being relieved from 40 minutes of lying supine on Dabir AP overlay as compared to that on regular OR overlay.

# Aim 3: To assess the feasibility of utilizing Dabir AP overlay for ischemic preconditioning for prolonged weight bearing condition.

**Hypothesis 3.** With 40 minutes of preconditioning using the Dabir AP overlay, our participants will demonstrate smaller reactive hyperemic response at sacrum and heel after being relieved from the regular OR overlay as compared to that without preconditioning.

#### 4.0 Eligibility

Twenty people with chronic SCI will be recruited from the Greater Chicago area. The eligibility of the subjects will be determined by the study team based on the following criteria.

#### 4.1 Inclusion Criteria

- Males and females 18-64 years old
- have had spinal cord injury for more than one year
- have injury level at T10 or above
- not ambulatory and use a wheelchair for mobility
- non smokers or able to refrain from smoking four hours prior to and during the study

#### 4.2 Exclusion Criteria

- current pressure ulcer
- history of diabetes mellitus
- history of cardiovascular diseases
- history of hypertension
- history of pulmonary diseases
- pregnant women (based on screening and pregnancy testing)
- non-English speakers

#### 4.3 Excluded or Vulnerable Populations

No vulnerable population will be included in the study. Since all key investigators are fluent only in English language, non-English speaking subjects will not be included.

#### 5.0 Subject Enrollment

Subjects will be eligible to participate in this study if they meet the study criteria as determined by the telephone screening and face-to-face screening procedures.

#### **Telephone Screening Procedure (approximately 15 minutes)**

Subjects will be recruited from the Greater Chicago area through study flyers. The PI or key personnel will recruit the eligible subjects when potential subjects call in response to the flyer. Questions regarding the inclusion and exclusion criteria will be asked to determine the eligibility based on the telephone screening script. Results of the telephone screening will be documented in Forms A, B, C1, C2, and D. If the potential subject is not eligible, results and confidential information will be destroyed immediately. All potential subjects will be scheduled to a study visit at the UIC Applied Health Sciences Building room 272 for further screening. Subjects will be asked to fast and refrain from smoking four hours prior to and during the study, and refrain from consuming any caffeinated foods/drinks for 12 hours prior to the study.

#### Face-to-face Screening Procedure (approximately 30 minutes)

Upon arrival for the study visit, the PI or key personnel will inform the potential subject of the study procedures and risks and benefits of the study. A consent form with details of all procedures, risks and benefits will be provided to the potential subject. Once the PI or key personnel receive the signed consent form, the subject will proceed to face-to-face screening. During the face-to-face screening procedure, the PI or key personnel will measure the resting heart rate and blood pressure with heart rate monitor and blood pressure cuff respectively and documented in form E1. The PI or key personnel will also examine the remaining motor function, sensation and autonomic function after spinal cord injury. The remaining sensation, motor, and autonomic function are standard physical examination for people with SCI in the clinic. The remaining sensation will be tested with the key personnel performing light touch of the skin below the level of injury (as the picture shown in form E2), and the motor function will be tested with the key personnel instructing subject to perform joint movement below the level of injury. Results of the remaining sensation and motor function will be documented in form E2. The autonomic function will be tested by asking subject questions regarding their ability to sweat, ability to sense the changes in temperature, bladder function, bowel movement and sexual function, and results will be documented in form E3. If the subject demonstrates normal heart rate and blood pressure, the subject will proceed with the study procedures. Women of childbearing age will also be screened for pregnancy using a urine pregnancy test strip. Women who are pregnant will not be eligible to participate.

#### 6.0 Study Design and Procedures

<u>Study Design</u>. This study uses a <u>repeated measures design</u>, and each subject will act as his/her own control. Each subject will undergo the two protocols in the experimental procedures: AP protocol and Control protocol. To ensure the order of the two protocols are randomized, the order of AP and Control protocols will be determined by drawing one envelope from the envelope pool. We will start with a pool of total 20 envelopes (10 envelopes indicating AP protocol first, and 10 envelopes indicating control protocol first). Once the envelope is drawn from the pool, it will not return to the pool.

<u>Study Procedures (Research purpose)</u>. After enrollment, subjects will proceed to the following procedures: 1) experimental procedures, 2) vascular control measures, 3) pressure mapping of wheelchair and 4) blood withdraw.

#### 1) Experimental procedure (approximately 4.5 hours)

Each subject will undergo two study protocols: AP and control (figure 1), and the order of the protocols will be randomized as described previously. A 30-minute washout period will be provided in between the two protocols. Two Laser Doppler flowmetry (LDF) flat probes (moor instrument, Wilmington, DE) will be taped to the sacrum and one heel to collect the skin blood flow response throughout both AP and control protocols. A whole body pressure mapping system (Xsensor, Xsensor Technology Corp., Alberta, Canada) will be used between the subject and the overlay to collect the inter pressure data. For the AP cycle, we will use four 10-minute cycles (5 minutes of high pressure and 5 minutes of low pressure).

<u>AP protocol:</u> The subject will first lie on his/her side quietly for 10 minutes to collect the baseline skin blood flow, followed by lying supine on the Dabir AP overlay for 40 minutes, and then side lying for 30 minutes to collect the first reactive hyperemic response. To test the effect of preconditioning, the subject will then lie supine on the OR overlay for 40 minutes followed by side lying for 30 minutes for the second reactive hyperemic response.

<u>Control protocol:</u> The subject will first lie on his/her side quietly for 10 minutes to collect the baseline skin blood flow, followed by lying supine on the OR overlay (AliMed®) for 40 minutes, and then side lying for 30 minutes to collect the reactive hyperemic response for control protocol.



Figure 1. Illustration of the full course of the experimental protocols: Alternating pressure (AP, top panel) and Control (Ctrl, bottom panel).

#### 2) Vascular control measures (approximately 30 minutes)

The PI, or key personnel will then collect the vascular control measures, including the <a href="heat hyperemic (HH) blood flow response">heat hyperemic (HH) blood flow response</a>, and the <a href="heat skin">skin</a> vasomotor response</a>. A non-invasive combined laser Doppler and white light reflectance spectroscopy (LDF-WLRS) probe (CP2T-1000, Moor Instrument, Wilmington, DE) will be used for both measures.

HH blood flow response will be measured at the sacrum and one heel while the subject is in side-lying position. Figure 2 demonstrates the HH measurement setting. HH will be induced with the heater at the tip of the probe head (41°C for 5 minutes). This HH measure will take approximately 7 minutes (2 min-baseline, 5 min-heating) per location. In total, the HH measures will take up to 15 minutes to complete.

The skin vasomotor response will be induced using cutaneous electrical stimulation (3-10 mA, 0.2-1.0 ms pulses at 20 Hz, 1 s trains) delivered via 1 cm Ag-AgCl surface electrodes applied bilaterally (4 cm apart) to the forehead (above lesion) and the abdominal wall (below lesion) while the subject is in a semi-reclined position. For each site, 5-8 stimuli will be delivered randomly. CP2T-1000 probe will be used to collect SBF and tissue oxygenation data at pulp of the second finger and toe. Subject will be in a semi-reclined position (about 30° from horizontal plane) during this protocol, and it will take up to 15 minutes to complete this protocol.



Figure 2. (A) hand held LDF-WLRS probe with heater ring, (B) HH measure.

#### 3) Pressure mapping of wheelchair (approximately 10 minutes)

The subject will be asked to transfer back to his/her wheelchair with the pressure mapping system placed between the wheelchair and the subject to collect the interface pressure data. The pressure mapping system is the same as that used between the subject and overlay to collect the interface pressure data.

#### 4) Blood withdraw (approximately 15 minutes)

The key personnel will draw venous blood samples (total 20 mL) via venipuncture for standard blood tests, including glycated hemoglobin (HbA1C), plasma glucose, lipid and lipoprotein concentrations (i.e. total-cholesterol, low-density lipoprotein, triglycerides, and high-density lipoprotein). The rationale for making these measurements is to collect potential covariates that might affect skin blood flow responses. Blood samples not used to probe for blood sugar and lipid profile tests will be stored up to five years (or until exhausted) for further analyses, since latest trend in literatures demonstrated metabolic syndrome after spinal cord injury had an effect on pressure ulcer formation.<sup>13</sup>

#### 7.0 Expected Risks/Benefits

#### **Expected Risks**

Overall, potential risks associated with participation in the study are unlikely and of low risk. Subjects will be advised to speak with the PI if they believe they have been hurt by the study. Potential risks associated with the non-invasive protocols of our study are as followed:

- <u>Emotional stress</u>: The risk of having emotional stress with our telephone screening procedure and examination of remaining sensation, motor and autonomic function is no more than minimal. Participants may feel uncomfortable answering personal health related questions. The examinations of remaining sensation, motor and autonomic function are regularly performed at the physician's office. Participants may feel uncomfortable that he or she could not feel or move the body below the level of injury. In addition, female subjects may feel added emotional stress if their screening pregnancy test results are positive and they were unaware that they were pregnant.
- <u>Oiscomfort:</u> The risk of having discomfort with our heart rate, blood pressure, exams is no more than minimal. These examinations are regularly performed at the physician's office. Participants may feel discomfort caused by the blood pressure cuff and heart rate monitor belt.
- 3) Localized Ischemia. The risk of tissue ischemia associated with reactive hyperemia (caused by lying on OR or AP overlays) is low. Reactive

hyperemia is a normal physiological response induced by short-term non-damaging ischemia of the loaded area. The amount of pressure expected on sacrum and heels is very low (~60mmHg) and for a short period of time (40 minutes), which simulates the amount of pressure lying or sitting on a mattress or seat cushion. The amount, duration and area of localized pressure on the skin is within the current clinical practice guideline of pressure ulcer prevention, which is making turning the patient in bed every two hours. The skin breakdown risk associated with lying on OR or AP overlay is considered as rare (less than 1 out of 100 people).

- 4) Localized Heating. The risk of burn associated with heat hyperemia is low. Heat hyperemia will be induced by short-term heating of the skin. The temperature of heating is very low (41°C or 106°F) and for a short period of time (5 minutes). This temperature and duration is far lower and shorter than the therapeutic hot packs used regularly in clinic (45-54°C) for more than 10 minutes covering the whole joint or lower back. Previous published literatures that investigated microcirculatory response in people with SCI induced heat hyperemia with 20-30 minutes heating at 41°C. No tissue burn or damage to the skin was noted in these published studies. The amount and duration of localized heating of the skin is far shorter than that causing burn of the skin. The skin breakdown risk associated with the heating protocol is considered as rare (less than 1 out of 100 people).
- <u>5)</u> Electrical Stimulation. The risk of skin or muscle damage associated with electrical stimulation is low. The skin vasomotor response will be induced using cutaneous electrical stimulation (3-10 mA, 0.2-1.0 ms pulses at 20 Hz, 1 s trains) delivered via 1 cm Ag-AgCl surface electrodes applied bilaterally (4 cm apart) to the forehead (above lesion) and the abdominal wall (below lesion). This is a standard protocol used to measure the sympathetic outflow of the microcirculatory response. The same protocol was used in previous studies on chronic spinal cord injury patients, and no damage to the skin or underlying muscle was noted. Electrical stimulation at a higher intensity and duration (10-50mA for 10 minutes) is one of the standard clinical practice protocol in nerve stimulation and pain reduction for patients with SCI. Therefore the skin or muscle damage associated with electrical stimulation is considered as rare (less than 1 out of 100 people).
- 6) Skin Blood Flow (SBF) and Tissue Oxygenation Testing will be performed using an FDA cleared non-invasive device. The amount of energy used with the laser light during the measurement is similar to that of a bar code scanner, and the white light is similar to that of ordinary daylight.
- 7) Bruising and swelling with venipuncture The risks of drawing blood from a vein includes discomfort at the site of the needle stick, possible bruising and swelling around the site of the needle stick is minimal. The risks of infection is very rare, and feeling faint from this procedure is uncommon.
- 8) Bare skin measurements. Bare skin measurements will be collected during this study. Some of the locations for the measurements, such as the sacrum

- (low back) is very private, so the subject may feel embarrassed. A bed sheet will be provided to cover the subjects upon request.
- <u>9)</u> Breach of confidentiality. The risk of breach of confidentiality is minimal since the only key to link subject ID and confidential information is locked in the file cabinet of the Pl's locked office. The key will only be accessible to the Pl's team. All other data is only coded with a subject ID in hard copy and electronic files. All hard copy files with subject ID only will be stored in a locked cabinet in the Pl's locked laboratory, which is three floors away from the Pl's office. All electronic data do not contain any confidential information, and they will be stored on the laptop used to collect data, and the hard drive located in the Pl's Laboratory. Both computers are password protected, and the data are only accessible to the Pl's team. All study personnel are trained in the maintenance of security and confidentiality of research data.

#### Benefits.

There is no direct benefit for the participants in this study, however findings from these participants will help us understand the potential benefit of the Dabir AP overlay as compared to the regular OR overlay, and the potential use of Dabir AP overlay on ischemia-preconditioning.

#### 8.0 Data Collection and Management Procedures

Three sets of data (and one biological sample) will be collected from the subjects. The following listed the details of data procurement, storage, and encryption: All data will be stored at UIC, and data will not be shared or stored at Schwab.

- 1) Confidential information (hard copy only): Confidential information that includes direct identifiers such as name, date of birth and phone number will be recorded on Form A. A subject ID (code) will be assigned to the subject by PI upon study enrollment for the purpose of protecting the confidentiality of the subject data for analysis purpose. Form A will serve as the key to the code. Form G is the compensation form. Participants will be asked to sign the form once the payment is received. Form A and G will be stored in a locked file cabinet in PI's locked office (UIC Applied Health Science Building, Rm 506H). Only the PI will have access to this locked file cabinet. A portable lock cash box will be used to transport Form A and G between the DHSP building and Department of Physical Therapy. Form A and G will be stored up to five years and destroyed afterwards so that all data will be de-identified for future analyses only.
- 2) Paper-based data (hard copy and excel spread sheet) will be coded using the subject ID on forms: B, C, D, E and F. These forms will be stored in a locked file cabinet in PI's locked laboratory (UIC Applied Health Science Building, Rm 272; different from the room that stores Forms A and G). The PI's team will be responsible for incorporating data on these forms to an excel

- spreadsheet for further statistical analyses. Two layers of encryption will be used to ensure the security of excel file. These coded data will be stored up to seven years after completion of this study.
- 3) Skin blood flow data (electronic text file generated automatically with data acquisition system): Skin blood flow data will be collected directly via the LDF. These analog signals are automatically stored on the UIC laptop used for data collection. Only Dr. Tzen's team can log on to the password protection laptop to collect and access the blood flow and tissue oxygenation data. The assigned subject ID will be the only identifier of the data set collected from each subject. These coded data will be stored up to seven years after completion of this study.
- 4) Blood sample: The blood samples not used to probe for blood glucose and lipid profile will be stored coded at co-investigator Dr. Haus' lab (UIC Applied Health Science Building, Rm 106). Dr. Haus will not have access to the key of the code.
- 5) Urine sample: Urine will be collected from women of childbearing age for pregnancy testing during visit one for eligibility screening. Any urine remaining after the testing will be disposed of.

#### 9.0 Data Analysis

The MatLab program (The MathWorks Natick, MA) will be used to process the skin blood flow signal. The signals will be analyzed with two signal processing methods to characterize the responses in both time and frequency domains. Details of both methods were published previously by the PI.<sup>14</sup>

- 1) Exponential curve-fitting technique:

  To select the time-domain parameters of the reactive hyperemia and heat hyperemia objectively. A tenth ordered Chebyshev I low pass filter (with cut off frequency at 0.15 Hz) will be applied to remove the noise caused by respiration and cardiac movement. We will use a least squares model to fit the filtered reactive and heat hyperemic curves, and all parameters (including peak, time to peak, area under curve of reactive hyperemia; and first peak, second peak and time to first and second peaks, area under curve of heat hyperemia) will be derived from the fit curves.
- 2) Time-frequency analysis:
  To further examine the different control mechanisms of SBF by decomposing the signal in frequency domain. Short-time Fourier transform will be used to decompose the signal by breaking the signal into short-time segments (windows), then computed Fourier analysis within each segment to calculate

spectral densities. A 256-sample Hanning window (512 seconds) will be used to compute the spectrogram.

Please see section 12.0 for details of all statistical analyses.

#### 10.0 Quality Control and Quality Assurance

Dr. Tzen will be responsible for quality control and quality assurance of the data collected. Dr. Tzen has more than ten years of experiences in pressure ulcer research using non-invasive blood flow measurements, and she will perform the protocols in person and shadow her research team on the first two subjects. Dr. Tzen will then supervise the data collection on site for the next three subjects recruited in this study. Dr. Tzen will check all the data within two days of collection (paper and electronic formats). If the study team encounter any issues related to data collection, Dr. Tzen is available through phone calls to address the concerns. Dr. Tzen will meet with her team every two weeks to check the laboratory notes and monitor the study regularly.

#### 11.0 Data and Safety Monitoring

The PI of this study (Tzen) will be responsible for monitoring the data and safety of this study. Dr. Tzen will meet with the research team every two weeks to monitor the overall conduct of the study (including issues with safety, ethics, recruitment, retention, adequacy of study design to achieve the specific aims) and provide feedback to the study team for the possible protocol amendments, and input from this study on future studies. Serious adverse events are not expected, but all such events will be reported according to the UIC IRB, and will be handled with the standard of Good Clinical Practice Guidelines including informing the PI, and IRB within 24 hours of the event, following up and reporting on the event until resolved, and subsequently reported to the PI.

The risk of breach of confidentiality is minimal since the only key to link subject ID and confidential information is a hard copy of Form A, which is locked in the file cabinet of the Pl's locked office. All other data is only coded with a subject ID in hard copy and electronic file. All hard copy files with subject ID only will be stored in a locked cabinet in the Pl's locked laboratory, which is three floors away from the Pl's office. All electronic data are also coded and encrypted using Symantec software, and they will be stored on the laptop used to collect data, and the hard drive located in the Pl's laboratory. Both computers are password protected, and the data are only accessible to the Pl's team. All study personnel are trained in the maintenance of security and confidentiality of research data.

#### 12.0 Statistical Considerations

For aims 1 and 2, paired *t*-tests will be computed to compare the interface pressure and skin blood flow during 40 minutes of AP overlay (AP protocol) vs. OR overlay (Ctrl protocol). Paired *t*-tests will also be used to compare the reactive hyperemic response during RH1 (AP protocol) vs. RH (Ctrl protocol). For aim 3, paired *t*-tests will be computed to compare the skin blood flow during OR overlay (AP protocol) vs. OR overlay (Ctrl protocol), and the reactive hyperemic response during RH2 (AP protocol) vs. RH (Ctrl protocol). SPSS will be used for all statistical analyses. Since this is a pilot study, we will test the study on 15 subjects. Results form this study will be used to calculate sample size for future studies. In case of dropout or subject decease during this study, we propose to recruit up to 20 subjects for this study.

#### 13.0 Regulatory Requirements

#### 13.1 Informed Consent

Oral consent will be obtained by phone during the initial telephone screen. Eligible subjects will be scheduled for a study visit where written informed consent will be obtained prior to conducting any study procedures. The PI's team is responsible for obtaining the signed consent form. The PI's team members were trained by the PI in obtaining informed consent, including thorough explanation of the research protocols and allowing potential subjects sufficient amount of time to ask any questions and to make the decision in participating in this study. To ensure the quality of the informed consent process, the PI will consent the first two subjects by herself and shadow her team members, and the PI will supervise her team members to consent the next three potential subjects of this study.

The informed consent documents will be stored in a locked file cabinet in PI's locked office (UIC Applied Health Science Building, Rm 506H), only the PI have access to the locked file cabinet. A portable lock cash box will be used to transport the signed consent forms from the DHSP building to the PI's office. Only the PI's team will have access to the consent form. Subjects will receive a signed copy.

#### 13.2 Subject Confidentiality

As described in 8.0 Data Collection and Management Procedures, the only document that contains confidential information is a hard copy of Forms A and G. To guard the confidentiality, Forms A and G will be stored in a locked file cabinet in PI's locked office (UIC Applied Health Science Building, Rm 506H), only the PI has access to this locked file cabinet. A portable lock cash box will be used to transport Form A between DHSP

building and the Pl's office. Form A and G will be destroyed at the end of the study so that all data will be de-identified for future analyses only.

Other data, including Forms B, C, D, E, F, blood flow and tissue oxygenation data in text files and excel spreadsheets will only contain an assigned subject ID, and Form A is the only document to link the subject ID to the subjects' confidential information. To guard the confidential information, Forms B, C, D, E, F will be stored in a locked file cabinet in Pl's locked laboratory (UIC Applied Health Science Building, Rm 272; different from the room that stores Forms A and G). The PI's team will be responsible for incorporating data on Form B to a excel spreadsheet that contains information of all subjects on a password protected desktop located in the PI's locked laboratory. Two layers of encryption will be used. The analog signals of blood flow and tissue oxygenation will be stored on the password protected UIC laptop used for data collection. Only the PI's team can access the laptop to collect and access data. The assigned subject ID will be the only identifier of the data set collected from each subject. These coded data will be stored up to seven years after completion of this study. The password of the laptop and desktop used in this study will be changed quarterly and known only by the PI's team.

#### 13.3 Unanticipated Problems

The PI will be responsible for monitoring and overseeing all procedures of the study. With the previous experiences, there should be no unanticipated problems with this study. However, should any unanticipated problems occur, the incident will be handled with the standard of Good Clinical Practice Guidelines including informing the PI, and IRB within 24 hours of the event, following up and reporting on the event until resolved, and subsequently reported to the PI.

#### 14.0 References

- 1. National Pressure Ulcer Advisory Panel. *Prevention and treatment of pressure ulcers: clinical practice guideline*. (2015).
- 2. HomeStar Meical Equipment & Infusion Services. Summary of medicare coverage for medical equipment.
- 3. Arias, S. *et al.* Effects on interface pressure and tissue oxygenation under ischial tuberosities during the application of an alternating cushion. *J. Tissue Viability* **24**, 91–101 (2015).
- 4. Jan, Y.-K., Brienza, D. M., Boninger, M. L. & Brenes, G. Comparison of skin perfusion response with alternating and constant pressures in people with spinal cord injury. *Spinal Cord* **49**, 136–141 (2011).
- 5. Masterson, S. & Younger, C. Using an alternating pressure mattress to offload heels in ICU. *Br. J. Nurs. Mark Allen Publ.* **23,** S44, S46–49 (2014).
- 6. Hausenloy, D. J. & Yellon, D. M. Remote ischaemic preconditioning: underlying mechanisms and clinical application. *Cardiovasc. Res.* **79**, 377–386 (2008).
- 7. Shaked, G. *et al.* Intermittent cycles of remote ischemic preconditioning augment diabetic foot ulcer healing. *Wound Repair Regen. Off. Publ. Wound Heal. Soc. Eur. Tissue Repair Soc.* **23**, 191–196 (2015).
- 8. Minson, C. T., Berry, L. T. & Joyner, M. J. Nitric oxide and neurally mediated regulation of skin blood flow during local heating. *J. Appl. Physiol. Bethesda Md* 1985 **91**, 1619–1626 (2001).
- 9. Nicotra, A., Asahina, M. & Mathias, C. J. Skin vasodilator response to local heating in human chronic spinal cord injury. *Eur. J. Neurol.* **11**, 835–837 (2004).
- 10. Tzen, Y.-T., Brienza, D. M., Karg, P. & Loughlin, P. Effects of local cooling on sacral skin perfusion response to pressure: implications for pressure ulcer prevention. *J. Tissue Viability* **19**, 86–97 (2010).
- 11. Nicotra, A., Young, T. M., Asahina, M. & Mathias, C. J. The effect of different physiological stimuli on skin vasomotor reflexes above and below the lesion in human chronic spinal cord injury. *Neurorehabil. Neural Repair* **19**, 325–331 (2005).
- 12. Brown, R., Engel, S., Wallin, B. G., Elam, M. & Macefield, V. Assessing the integrity of sympathetic pathways in spinal cord injury. *Auton. Neurosci. Basic Clin.* **134**, 61–68 (2007).
- 13. Li, C., DiPiro, N. D., Cao, Y., Szlachcic, Y. & Krause, J. The association between metabolic syndrome and pressure ulcers among individuals living with spinal cord injury. *Spinal Cord* **54**, 967–972 (2016).
- 14. Tzen, Y.-T., Brienza, D. M., Karg, P. E. & Loughlin, P. J. Effectiveness of local cooling for enhancing tissue ischemia tolerance in people with spinal cord injury. *J. Spinal Cord Med.* **36**, 357–364 (2013).

#### **APPENDICES**

### American Spinal Injury Association (ASIA) Impairment Scale

A = Complete: No motor or sensory function is preserved in the sacral segments S4-S5.

B = Incomplete: Sensory but not motor function is preserved below the neurological level and includes the sacral segments S4-S5.

C = Incomplete: Motor function is preserved below the neurological level, and more than half of key muscles below the neurological level have a muscle grade less than 3.

D = Incomplete: Motor function is preserved below the neurological level, and at least half of key muscles below the neurological level have a muscle grade of 3 or more.

E = Normal: motor and sensory function are normal.

| Dabir AP Overlay (PI: Tzen): Alternating Pressure Overlay on Weight Bearing Tissue Tolerance in So | Cl |
|---|---|
| Research Data Collection Forms | |
| Subject ID: | |

# **FORM A: CONFIDENTIAL INFO**

| Name of subject: | | | |
|------------------------|--------|---|--------------|
| Date of birth:// | | | |
| Address: | | | |
| Street: | | | |
| City: | State: | | Zip Code: |
| E-mail: | | | |
| | | Г | |
| | | | IRB approval |
| | | L | |
| Researcher's Initials: | | | |
| Date: | | | |

| Dabir AP Overlay (PI: Tzen): Alternating Pressure Overlay on Weight Bearing Tissue Tolerance in So | Cl |
|---|---|
| Research Data Collection Forms | |
| Subject ID: | |

# FORM B: DEMOGRAPHIC INFO

| Gender: Male Female | |
|---|---|
| <ul><li>Weight: Height:</li><li>(Body Mass Index:</li></ul> | (To be calculated by the investigator) |
| Race/Origin:African-American | Asian-American/Asian |
| Caucasian | Hispanic |
| Others (please specify | ) |
| | IRB approval |

| Dabir AP Overlay (PI: Tzen): Alternating Pressure Overlay on Weight Bearing Tissue Tolerance in S | CI |
|---|---|
| Research Data Collection Forms | |
| Subject ID: | |

# **FORM C1 – SELF-REPORT MEDICAL HISTORY**

| Spinal Cord Injury History | |
|---|---|
| • Date of injury:/ | |
| • Level of injury: Cervical Thoracic Lumbar_ | |
| • AIS: A B C | |
| Wheelchair: manual power | |
| Pregnant: yes no | |
| Other Medical history | IRB approval |
| Cardiovascular Disease | |
| Hypertension | |
| Diabetes Mellitus | |
| Neuropathy | |
| Lung Disease | |
| Others, please list | |
| None of above diseases | |
| Pressure Ulcer history | |
| If had pressure ulcers in the past, please indicate the le | ocation and time: |

| Dabir AP Overlay (PI: Tzen): Alternating Pressure Overlay on Weight Bearing Tissue Tolerance in SC |
|---|
| Research Data Collection Forms |
| Subject ID: |

# **FORM C2 – SELF-REPORT CURRENT MEDICATION**

| Name of Medication | Dosage | Frequency | Reason for Taking |
|--------------------|--------|-----------|-------------------|
| | | | IRB approval |

| Dabir AP Overlay (PI: Tzen): Alternating Pressure Overlay on Weight Bearing Tissue Tolerance in So | CI |
|---|---|
| Research Data Collection Forms | |
| Subject ID: | |

# FORM D - SELF-REPORT SOCIAL HISTORY

| Please indicate <u>Yes</u> or <u>No</u> to the following: Do you smoke?YesNo | |
|---|---|
| If yes, packs per day? | Number of years? |
| Do you exercise on a regular basis?Yes _<br>If yes, describe | |
| | IRB approval |
| Researcher's Initials: | |

| Research Data Collection Form | | Ŭ |
|-------------------------------|--------------------|-------|
| Subject ID: | _ | |
| FC | DRM E1 _ RESTING V | PIATI |

(to complete during face-to-face screening)

| Resting heart ra | ate: | |
|------------------|-----------|---------------------------------|
| Resting blood p | oressure: | |
| Pregnant: | yes | no (based on urine test result) |

#### FORM E2 - ASIA IMPAIRMENT SCALE

(to complete during face-to-face screening)



# Muscle Function Grading

- 1 = palpable or visible contraction
- 2 = active movement, full range of motion (ROM) with gravity diminated
  - 3 = active movement, tul ROM against gravity
- 4 = active movement, till ROM against gravity and moderate resistence in a muscle specific position

B = Sensory Incomplete. Sensory but not motor function is preserved below the reundogical level and includes the social

A = Complete. No sensory or motor function is preserved in

the sacral segments S4-5.

4SIA Impairment Scale (AIS)

 $\mathbf{5}^+$  = (normal) active movement, LLI ROM against grawly and sufficient resistance to be considered normal if identified inhibiting factors (i.e. pah., deuse) were not present 5= (roma), active movement. UI ROM against gravity and UII resistance in a tradicial muscle position expected from an ofnewise unimpared person

NT = not estable (i.e. due to immobilizaton, severe pain such that the patient carnot be graded, amputation of limb, or contracture of > 50% of the normal ROM)

# Sensory Grading

- = Altered, either decreased/impaired sensation or hypersensitivity
  - 2 = Normal
    - NT = Not testable

# When to Test Non-Key Muscles:

In a patient with an apparent AIS B classification, non-key muscle functions more than 3 leads below the mofor beloi on each side should be tested to most accurate classific the intimor infinementals between AIS R and Ct

D = Motor Incomplete, Motor incomplete status as defined

above, with at least half that for more) of hey muscle functions

celow the single NU having a muscle grade ≥ 3.

E = Normal. If sensation and motor tunction as tested with

the ISNOSCI are graded as normal in all segments, and the patenthad prior delicits, then the AIS grade is E. Someone

without an initial SCI does not receive an 4IS grade.

musde functions below the single NU have a muscle grade ≥ 3.

| Movement Root let | Root level |
|-------------------------------------------------------------|------------|
| Shoulder: Revion, extension, abduction, adduction, internal | 용 |

| Movement | HOOF BYE |
|---|---|
| Shoulder: Pexion, extension, abduction, adduction, internal and external rotation<br>Elbow: Sugination | 용 |
| Elbow: Proraton<br>Wrist: Rexon | 8 |
| Finger: Reaton at proximal joint, extension.<br>Thumb: Reaton, extension and abolicion in plane of frumb | CJ |
| Finger: RevionatMOP joint Thumb: Opposition, adduction and adduction perpendicular to palm | පී |

| Finger, Abduction of the inclay linger | H |
|--------------------------------------------------------------|----|
| Hip: Adduction | 71 |
| Hip: External rotation | 23 |
| Hip: Extension, abduction, internal notation<br>More playing | 14 |
| Ankle: Inversion and eversion | |

# INTERNATIONAL STANDARDS FOR NEUROLOGICAL CLASSIFICATION OF SPINAL CORD INJURY ध ह Hallux and Toe: DP and RIP flexion and abouncion

Toe: MP and Pedersion

# Steps in Classification

The following order is recommended for determining the dassification of ndviduals with SQ.

- The sansary lard is the most causal, idact damatome for both pin prick and Determine sensory levels for right and left sides. light fourth sensetion.
- aresumed to be the same as the sensory level, if testable motor function above supine testing), providing the key muscle fundions nearesented by segments Defined by the lowest key muscle function that has a grade of at least 3 (on above that lavel are jodged to be infact (graded as a S). Note: in regions where there is no myotome to test, the motor lavel is Determine motor levels for right and left sides. that level is also normal.

most caudal sacral segments for voluntary anal contraction (VAC)

C = Motor Incomplete. Motor function is preserved at the

pressure) AND no motor function is preserved more than three levels below the motor level on either side of the body.

segments S4-5 (light buch or pinpiick at S4-5 or deep anal

(sensory function preserved at the most caudal sacral segments

(\$4.85) by LT, PP or DAP), and has some spaning of motor

OR the patient meets the criteria for sensory incomplete status

function more than three levels below the ipsilateral motor level

(This includes key or non-key musdle functions to determine

on either side of the body.

notor incomplete status.) For AIS C - less tranhalf of key

- antigravity (3 ormore) muscle function strength, provided that there is norma (inted) sensay and molar function rostally respectively. The NLI is the most ceptalled of the sensay and molar levels determined in This refers to the most cautal segment of the cord with intact sensation and 3. Determine the neurological level of injury (NLI) steps 1 and 2.
- If volutary anal contraction = No AND all S4-5 sensory scores = 0 Determine whether the injury is Complete or Incomplete. AND deep anal pressure = Mg, then injury is Compliate (i.e. absence or presence of sacral sparing) Otherwise, irjuny is Incomplete.
- If YES, AIS = A and can record 5. Determine ASIA Impairment Scale (AIS) Grade: Is injury Complete?



Using ND: To document the sensory, motor and NLI levels,

the ASIA Impairment Scale grade, and/or the zone of partal

preservation (279) when hey are unable to be determined based on the examination results.



are at least half (half or more) of the key muscles below the <u>neurological</u> level of injury graded 3 or better?



If sensation and motor function is normal in all segments, AIS=E.
Note: AIS E is used in follow-up lesting when an individual with a document of
SCI has recovered normal function. If all initial lesting no delicitis are found, the individual is neurologically infact, the ASIA Impairment Scale does not apply



Hallux: Adduction

| Dabir AP Overlay (PI: Tzen): Alternating Pressure Overlay on Weight Bearing Tissue Tolerance in SCI |
|---|
| Research Data Collection Forms |
| Subject ID: |

# **FORM E3 – AUTONOMIC FUNCTION SCALE**

| Manif | | - |
|------------|----------------|-------------|
| AMERICANIA | DINIAL INDUIDA | ASSOCIATION |



| Patient Name:<br>(Doo<br><b>General Auto</b> r | | ubject ID instead) | | Autonomic Diagnosis: (Supraconal □, Conal □, Cauda Equi <b>Lower Urinary Tract, Bowel and Sexual Function</b> | |
|---|---|---|---|---|---|
| System/Organ | Findings | | Check<br>mark | System/Organ | Score |
| Autonomic | Normal | | | Lower Urinary Tract | |
| control of the | Abnormal | Bradycardia | | Awareness of the need to empty the bladder | |
| heart | | Tachycardia | | | |
| | | Other dysrhythmias | | Ability to prevent leakage (continence) | |
| | Unknown | | | Bladder emptying method (specify) | |
| | Unable to assess | | | Bowel | |
| Autonomic | Normal | | | Sensation of need for a bowel movement | |
| control of<br>blood | Abnormal | Resting systolic blood pressure below 90 mmHg | | Ability to Prevent Stool Leakage (continence) | |
| pressure | | Orthostatic hypotension | | Voluntary enhinctor contraction | |
| | | Autonomic dysreflexia | | Voluntary sphincter contraction | |
| | Unknown | | | Sexual Function | |
| | Unable to assess | | | Genital arousal (erection or lubrication) Psychogenic | |
| Autonomic | Normal | | | Reflex | |
| control of sweating | Abnormal | Hyperhydrosis above lesion | | | |
| Sweating | | Hyperhydrosis below lesion | | Orgasm | |
| | | Hypohydrosis below lesion | - | Ejaculation (male only) | |
| | Unknown | | | | |
| | Unable to assess | | | Sensation of Menses (female only) | |
| Temperature | Normal | | | 2=Normal function, 1=Reduced or Altered Neurological Fun | nction |
| regulations | Abnormal | Hyperthermia | | 0=Complete loss of control, NT=Unable to assess due to preed concomitant problems | |
| | | Hypothermia | | | |
| | Unknown | | | | |
| | Unable to assess | | | | |
| Autonomic and | Normal | | | | |
| Somatic Control<br>of Broncho-<br>pulmonary<br>System | Abnormal | Unable to voluntarily breathe requiring full ventilatory support | | Date of Injury Date of Assessment | |
| | Impaired voluntary breathing requiring partial vent support | | | This form may be freely copied and reproduced but not modified. This assessment should use the terminology found in the Internation | |
| | | Voluntary respiration impaired does not require vent support | | SCI Data Sets (ASIA and ISCoS - http://www.iscos.org.uk) | |
| | Unknown | | | | |
| | Unable to | | | Evaminar | |

| Dabir AP Overlay (PI: Tzen): Alternating Pressure Overlay on Weight Bearing Tissue Tolerance in SCI |
|---|
| Research Data Collection Forms |
| Subject ID: |
| • |

### FORM F - TEST DATA

Envelope A: CTRL → AP

| Session | Heart Rate | Blood Pressure | |
|---------|--------------|----------------|-------|
| | Before After | Before | After |
| CTRL | | | |
| AP | | | |

Envelope B: AP → CTRL

| Session | Heart Rate | Blood Pressure | |
|---------|--------------|----------------|-------|
| | Before After | Before | After |
| AP | | | |
| CTRL | | | |

| (Signature of Investigator) | (Date) |
|-----------------------------|--------|

| Dabir AP Overlay (PI: Tzen): Alternating Pressure Overlay on Weight Bearing Tissue Tolerance Research Data Collection Forms Subject ID: | | | |
|---|---|---|---|
| FORM G – COMPEN | SATION | | |
| | edge that I am to | receive | |
| compensation for participating in this study \$ | on | / | / |

Researcher's signature \_\_\_\_\_\_Date\_\_\_\_